CLINICAL TRIAL: NCT00256139
Title: CLEAR Study: Clinical Experience Acquired With Raptiva Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24011
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Moderate to Severe Psoriasis
MeSH Terms: interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva

SUMMARY:
A multicentre, randomised, double blind, placebo controlled phase III study of subcutaneously administered Raptiva in the treatment of patients with moderate to severe psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Plaque psoriasis covering ³10% of total BSA (see Appendix A)
* Diagnosis of psoriasis for at least 6 months
* A minimum PASI score of 12.0 at screening (see Appendix A)
* Patients who are either not controlled by, intolerant to or contraindicated to at least 2 currently available systemic therapies (e.g., photochemotherapy (PUVA), cyclosporin, corticosteroids, methotrexate, oral retinoids, MMF, thioguanine, hydroxyurea, sirolimus, azathioprine, 6 MP) (defined as "high need" patients)
* Body weight <= £120 kg
* 18 to 75 years old
* For women of childbearing potential, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources during the study
* Willingness to enter Study

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* History of severe allergic or anaphylactic reactions to humanised monoclonal antibodies or fusion proteins that contain an Ig Fc region
* Clinically significant psoriasis flare during screening or at the time of enrollment
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV) Patients will undergo mandatory testing at screening. Patients who are positive for HIV will be excluded.
* Pregnancy or lactation
* WBC count <4000/mL or >14,000/mL
* Seropositivity for hepatitis B or C virus Patients will undergo testing during screening. Patients who are positive for hepatitis B antigen or hepatitis C antibody will be excluded.
* Hepatic enzymes ³3 times the upper limit of normal
* History of active tuberculosis (TB) or currently undergoing treatment for TB PPD testing or chest X-ray is required for high risk patients (see Appendix I). Patients with a positive PPD (not due to BCG vaccination) or chest X-ray will be excluded.
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders Patients with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled.
* Previous treatment with Raptiva (anti-CD11a)
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Serum creatinine ³2 times the upper limit of normal
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* History of substance abuse within the last 5 years
* Any medical condition that, in the judgment of the investigator, would jeopardize the patient's safety following exposure to study drug

Note: Restrictions and/or directions apply to the following treatments during specified time periods prior to initial study drug administration and during the study:

* Systemic therapy for psoriasis (within 28 days prior to Study Day 0)
* Systemic immunosuppressive drugs for other indications (within 28 days prior to Study Day 0)
* Topical therapies for psoriasis (within 14 days prior to Study Day 0)
* Live or killed virus or bacteria vaccines (within 14 days prior to Study Day 0)
* Other vaccines or allergy desensitisation (it is recommended that these are scheduled at least 14 days prior to Day 0 or ³3 months after the last injection of study drug)
* Other experimental drugs or treatments (within 28 days or five half lives, whichever is longer, prior to Day 0) b Blockers, ACE inhibitors, interferons, quinidine, antimalarial drugs, or lithium (if clinically indicated, such medications are allowed but the dosage should be held constant from Day -28 throughout the study)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2003-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Natta, M.D., Study Director — Sponsor GmbH
Locations (1):
- Serono International SA, Geneva, Switzerland

REFERENCES:
- [Result] Dubertret L, Sterry W, Bos JD, Chimenti S, Shumack S, Larsen CG, Shear NH, Papp KA; CLEAR Multinational Study Group. CLinical experience acquired with the efalizumab (Raptiva) (CLEAR) trial in patients with moderate-to-severe plaque psoriasis: results from a phase III international randomized, placebo-controlled trial. Br J Dermatol. 2006 Jul;155(1):170-81. doi: 10.1111/j.1365-2133.2006.07344.x. PMID 16792770
- [Derived] Ortonne JP, Shear N, Shumack S, Henninger E; CLEAR Multinational Study Group. Impact of efalizumab on patient-reported outcomes in high-need psoriasis patients: results of the international, randomized, placebo-controlled Phase III Clinical Experience Acquired with Raptiva (CLEAR) trial [NCT00256139]. BMC Dermatol. 2005 Dec 16;5:13. doi: 10.1186/1471-5945-5-13. PMID 16359548
- See also: CLEAR trial — http://www.biomedcentral.com/1471-5945/5/13